CLINICAL TRIAL: NCT06665230
Title: A Three-Period Study to Evaluate the Effects of Modafinil on the Single-Dose Pharmacokinetics of MK-6552 in Healthy Male Participants
Brief Title: A Clinical Study of MK-6552 and Modafinil in Healthy Men (MK-6552-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6552-005; MK-6552-005 (Other: MSD)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-6552 + Modafinil (Experimental): In Period 1, participants receive MK-6552 orally. In Period 2, participants receive MK-6552 orally plus low dose modafinil orally. In Period 3, participants receive MK-6552 orally plus high dose modafinil orally.
  Interventions: Drug: MK-6552; Drug: Modafinil

INTERVENTIONS:
Drug: MK-6552 — Oral administration
Drug: Modafinil — Oral administration
  Other Names: Provigil®

SUMMARY:
The goal of this study is to learn what happens to MK-6552 in a person's body over time. Researchers will compare what happens to levels of MK-6552 in people's blood when it is taken with and without modafinil. Researchers also want to learn about the safety of MK-6552 taken with and without modafinil and if people tolerate it.

ELIGIBILITY:
Inclusion Criteria

The main inclusion criteria include but are not limited to the following:

* Is in good health based on medical history and physical examination
* Has a body mass index ≥18 and ≤32 kg/m^2, inclusive

Exclusion Criteria

The main exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 1 month
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 19 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
High Dose Modafinil Effect: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-inf) of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the AUC0-inf of MK-6552 in the presence of high dose modafinil.
High Dose Modafinil Effect: Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of MK-6552 | At designated timepoints (up to approximately 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24hrs of MK-6552 in the presence of high dose modafinil.
High Dose Modafinil Effect: Time to Maximum Plasma Concentration (Tmax) of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the Tmax of MK-6552 in the presence of high dose modafinil.
High Dose Modafinil Effect: Maximum Plasma Concentration (Cmax) of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the Cmax of MK-6552 in the presence of high dose modafinil.
High Dose Modafinil Effect: Plasma Concentration of MK-6552 at 6 Hours Postdose (C6hrs) | At designated timepoints (up to approximately 6 hours postdose)
  Blood samples will be collected to determine the C6hrs of MK-6552 in the presence of high dose modafinil.
High Dose Modafinil Effect: Plasma Concentration of MK-6552 at 8 Hours Postdose (C8hrs) | At designated timepoints (up to approximately 8 hours postdose)
  Blood samples will be collected to determine the C8hrs of MK-6552 in the presence of high dose modafinil
High Dose Modafinil Effect: Apparent Clearance (CL/F) of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the CL/F of MK-6552 in the presence of high dose modafinil.
High Dose Modafinil Effect: Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the Vz/F of MK-6552 in the presence of high dose modafinil.
High Dose Modafinil Effect: Apparent Terminal Half-life (t1/2) of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the t1/2 of MK-6552 in the presence of high dose modafinil.

SECONDARY OUTCOMES:
Low Dose Modafinil Effect: AUC0-inf of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the AUC0-inf of MK-6552 in the presence of low dose modafinil.
Low Dose Modafinil Effect: AUC0-24hrs of MK-6552 | At designated timepoints (up to approximately 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24hrs of MK-6552 in the presence of low dose modafinil.
Low Dose Modafinil Effect: Tmax of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the Tmax of MK-6552 in the presence of low dose modafinil.
Low Dose Modafinil Effect: Cmax of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the Cmax of MK-6552 in the presence of low dose modafinil.
Low Dose Modafinil Effect: C6hrs of MK-6552 | At designated timepoints (up to approximately 6 hours postdose)
  Blood samples will be collected to determine the C6hrs of MK-6552 in the presence of low dose modafinil.
Low Dose Modafinil Effect: C8hrs of MK-6552 | At designated timepoints (up to approximately 8 hours postdose)
  Blood samples will be collected to determine the C8hrs of MK-6552 in the presence of low dose modafinil.
Low Dose Modafinil Effect: CL/F of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the CL/F of MK-6552 in the presence of low dose modafinil.
Low Dose Modafinil Effect: Vz/F of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the Vz/F of MK-6552 in the presence of low dose modafinil.
Low Dose Modafinil Effect: t1/2 of MK-6552 | At designated timepoints (up to approximately 36 hours postdose)
  Blood samples will be collected to determine the t1/2 of MK-6552 in the presence of low dose modafinil.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Alliance for Multispecialty Research, LLC (Site 0001), Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com